CLINICAL TRIAL: NCT00792935
Title: A Phase IIa, Multicenter, Double-Blind, Randomized, Active-Controlled, Parallel-Arm Clinical Trial to Study the Efficacy and Safety of MK-0941 Compared to Sulfonylurea in Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin Therapy
Brief Title: A Study to Test MK-0941 in Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin (MK-0941-017)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0941-017; 2008_589; CTRI/2009/091/000154 (Registry Identifier: CTRI)
Record Dates: First submitted 2008-11-14; First posted 2008-11-18 (Estimated); Results first posted 2012-10-03 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-((6-(ethylsulfonyl)-3-pyridinyl)oxy)-5-(2-hydroxy-1-methylethoxy)-N-(1-methyl-1H-pyrazol-3-yl)benzamide; glimepiride; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MK-0941 (Experimental)
  Interventions: Drug: MK-0941; Drug: Metformin
- Glimepiride (Active Comparator)
  Interventions: Drug: Glimepiride; Drug: Metformin

INTERVENTIONS:
Drug: MK-0941 — MK-0941 will be taken three times a day (TID), within 15 minutes before each meal. MK-0941 will be titrated to a maximally effective dose. The treatment period will be 6 weeks.
  Arms: MK-0941
Drug: Glimepiride — Glimepiride will be taken once a day (QD) in the morning, within 15 minutes before the breakfast meal. Glimepiride will be titrated to a maximally effective dose. The treatment period is 6 weeks.
  Other Names: Amaryl®
  Arms: Glimepiride
Drug: Metformin — The study will include an up to 4-week metformin dose titration/dose stabilization period. Once a participant has reached the maximum tolerated dose of metformin [(i.e., ≥1500 mg/day and ≤2550 mg/day (or ≤3000 mg/day, where the maximum dose of metformin per the local label is 3000 mg/day)], the participant should remain on the same metformin dose throughout the study.

SUMMARY:
The purpose of this study is to test the effect of MK-0941 as add-on therapy for participants taking metformin for type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patient has type 2 diabetes mellitus
* Between the ages of 18 and 70

Exclusion Criteria:

* Patient has a history of type 1 diabetes mellitus or ketoacidosis.
* Patient is on a weight loss program and is not in the maintenance phase or is taking weight loss medication.
* Patient has had surgery within 30 days of starting the study or has planned major surgery during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-0941: Participants receive MK-0941 5 mg or 10 mg tablets, orally, TID and placebo tablets matching glimepiride 1 mg or 2 mg, orally, QD for 6 weeks. Up-titration and down-titration of the dose could occur to achieve optimal individual glucose control. In addition, all participants received a maximum tolerated dose of metformin [(i.e., ≥1500 mg/day and ≤2550 mg/day (or ≤3000 mg/day, where the maximum dose of metformin per the local label is 3000 mg/day)], after a 4-week dose titration/dose stabilization period.
- Glimepiride: Participants receive glimepiride 1 mg or 2 mg tablets, orally, QD and placebo tablets matching MK-0941 5 mg or 10 mg, orally, TID for 6 weeks. Up-titration and down-titration of the dose could occur to achieve optimal individual glucose control. In addition, all participants received a maximum tolerated dose of metformin [(i.e., ≥1500 mg/day and ≤2550 mg/day (or ≤3000 mg/day, where the maximum dose of metformin per the local label is 3000 mg/day)], after a 4-week dose titration/dose stabilization period.
Period: Overall Study
Arm/Group | MK-0941 | Glimepiride
Started | 72 | 71
Completed | 68 | 68
Not Completed | 4 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0941 | Glimepiride | Total
Number analyzed (Participants) | 72 | 71 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (9.5) | 55.2 (9.8) | 55 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 43 | 45 | 88
Mean 24-Hour Weighted Mean Glucose at Baseline [Mean (Standard Deviation); unit: mg/dL] — Weighted Mean Glucose (WMG) is a measure of the amount of glucose in the blood over a period of 24 hours. The WMG was derived from multiple glucose values collected during both fasting and post-meal periods. The "weighted" mean was used to avoid over-representation of post-meal glucose values.
  mg/dL | 178.8 (33.9) | 184.4 (38.4) | 181.6 (36.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in 24-hour Weighted Mean Glucose
Description: Weighted Mean Glucose (WMG) is a measure of the amount of glucose in the blood over a period of 24 hours. The WMG was derived from multiple glucose values collected during both fasting and post-meal periods. The "weighted" mean was used to avoid over-representation of post-meal glucose values.
Time Frame: Baseline and Week 6
Population: The full analysis set (FAS) population included all randomized participants who had efficacy measurements at baseline or a post-randomization visit).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MK-0941 | Glimepiride
Number analyzed (Participants) | 72 | 71
mg/dL | -43.4 [-50.0 to -36.8] | -44.2 [-50.9 to -37.5]
Statistical Analysis 1: Comparison: MK-0941 vs Glimepiride; Using a standard deviation of 23.5 mg/dL, a sample size of at least 65 participants per treatment group would be required to have an 80% power to detect a true difference of 12.5 mg/dL between MK-0941 and glimepiride as measured by change from baseline in 24-hour WMG at Week 6; Test type: Superiority or Other; p = 0.847, Constrained longitudinal analysis; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-7.9 to 9.6], Standard Error of Mean 4.4

2. Primary Outcome: Number of Participants Who Experienced One or More Episodes of Hypoglycemia (Symptomatic or Asymptomatic)
Description: Hypoglycemic episodes are defined as either a fingerstick glucose
  measurement of ≤70 mg/dL [3.9 mmol/L] with or without symptoms or symptomatic hypoglycemia.
Time Frame: Baseline to Week 6
Population: All patients as treated (APaT) defined as all randomized participants who received at least one dose of MK-0941 or glimepiride.
Measure: Number; unit: participants
Arm/Group | MK-0941 | Glimepiride
Number analyzed (Participants) | 72 | 71
participants | 32 | 37
Statistical Analysis 1: Comparison: MK-0941 vs Glimepiride; Test type: Superiority or Other; p = 0.361, Miettinen & Nurminen method; Proportions = -7.7, 95% CI 2-sided [-23.6 to 8.7] — The estimated value represents the difference in percentages, MK-0941 minus Glimepiride

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: All randomized participants who received at least one dose of MK-0941 or glimepiride. Assessments during regular visits to the site (every 2 to 4 weeks).
Groups:
- MK-0941: All patients as treated (APaT) defined as all randomized participants who received at least one dose of MK-0941.
- Glimepiride: All patients as treated (APaT) defined as all randomized participants who received at least one dose of glimepiride.
Arm/Group | MK-0941 | Glimepiride
Serious Adverse Events (participants affected / at risk) | 1/72 | 1/71
Other Adverse Events (participants affected / at risk) | 31/72 | 25/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0941 (N=72) | Glimepiride (N=71)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0941 (N=72) | Glimepiride (N=71)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 28 (89) | 23 (78)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.